CLINICAL TRIAL: NCT05812482
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Safety and Efficacy of Urethral Drug Balloon Catheter in the Treatment of Urethral Stricture
Brief Title: Treatment of Urethral Stricture With Urethral Drug Ball
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPCTP-2021-009
Record Dates: First submitted 2023-03-15; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-08

CONDITIONS: Urethral Stricture Less Than 2 cm
Keywords: Urethral stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The test arm will be the treated by Drug Balloon
  Interventions: Procedure: Drug balloon dilatation
- Control group (Other): The control arm will be treated by Direct vision internal urethrotomy (DVIU)
  Interventions: Procedure: Direct vision internal urethrotomy (DVIU)

INTERVENTIONS:
Procedure: Drug balloon dilatation — The Drug balloon is covered with paclitaxel coating that diffuses the drug into the urethral wall when dilated
  Arms: Test group
Procedure: Direct vision internal urethrotomy (DVIU) — A control subject will choose DVIU surgery until the desired effect is achieved
  Arms: Control group

SUMMARY:
To evaluate the safety and efficacy of urethral drug balloon catheter in the treatment of urethral stricture.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled, and superiority study. The two groups were randomly selected into a total of 150 subjects (75 in the test group and 75 in the control group) according to 1:1. The test group was treated with urethral drug balloon catheter from Lepu Medical Technology (Beijing) Co.,Ltd., while the control group was treated with direct vision internal urethrotomy (DVIU).

All subjects were followed up at 1, 3 and 6 months post-procedure, and the efficacy of urethral drug balloon catheter will be evaluated with the success rate of operation at 6 months as the main end point. Observe the occurrence of complications and other indicators to make a reliable evaluation of the safety of urethral drug balloon catheter.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 and ≤ 85 years old, male patients;

  2. Urethral stricture was confirmed by transurethral angiography, and the length of stricture was less than 2 cm;

  3. Maximum urine flow rate (Qmax)<15 ml/s;

  4. There are obvious symptoms of urinary tract stricture such as slow urine rheology, difficulty in urination and incomplete urination;

  5. International Prostate Symptom Score (IPSS) ≥ 13;

  6. The guide wire must be able to pass through the stenosis segment;

  7. Patients who can understand the purpose of the trial, voluntarily participate in and sign the informed consent form, can independently complete effective questionnaires, and are willing to conduct clinical follow-up according to the research requirements.

Exclusion Criteria:

* 1. Patients with multiple stenotic lesions;

  2. Patients with a history of allergy to paclitaxel and contrast agents, or patients undergoing treatment with drugs that may antagonize paclitaxel;

  3. Patients who have undergone hypospadias repair, urethroplasty, stricture expansion or incision in the past 3 months;

  4. Urethral stricture caused by the following causes: bacterial urethritis, untreated gonorrhea, lichen sclerosus or dry glans obliterans;

  5. There are other diseases that can cause lower urinary tract symptoms, such as overactivity of bladder, neurogenic bladder dysfunction, etc;

  6. There are adverse factors for catheter insertion;

  7. Patients with artificial penis or urethral sphincter, or urethral or prostate stent;

  8. Patients who have been diagnosed with urethra cancer, bladder cancer cancer or prostate cancer, or who have experienced pelvic radiotherapy in the past 2 years;

  9. For patients with severe renal insufficiency, their serum creatinine is more than 2.5mg/dL or they are undergoing hemodialysis;

  10. Patients with severe lung disease, cardiovascular disease, coagulation dysfunction and contraindication of anesthesia;

  11. Patients with poor control of diabetes (hemoglobin A1c>8.0%);

  12. Patients with active urinary stones in the past 6 months;

  13. Patients who are not suitable for direct vision internal urethrotomy;

  14. Patients with pregnancy preparation plan;

  15. Patients who are participating in clinical trials of other drugs or medical devices and have not reached their main endpoint;

  16. Patients who cannot participate in the clinical trial due to other reasons considered by the investigator.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 6 months post-procedure
  no reoperation or instrument intervention is required, and 16F bladder flexible mirror or 16F catheter can pass through the stenosis

SECONDARY OUTCOMES:
Change in the International Prostate Symptom Score (IPSS) | 1, 3 and 6months
Change in the Quality of life index score (QOL) | 1, 3 and 6months
Maximum urinary flow rate (Qmax) | 1 and 6 months post-procedure
Residual urine volume (PVR) | 6 months post-procedure
Postoperative complications | 1,3,6 months post-procedure
  bleeding, false passage formation, rectal injury, infection, etc
Number of re-interventions after operation | 1, 3, 6 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jianbing Li, Study Director — Beijing Tsinghua Changgeng Hospital; Jianbin Bi, Study Director — First Hospital of China Medical University; Qiang Fu, Study Director — Shanghai 6th People's Hospital; Shaogang Wang, Study Director — Tongji Hospital affiliated to Tongji Medical College HUST; Xiaoping Zhang, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Yuanjie Niu, Study Director — Tianjin Medical University Second Hospital; Jinjian Yang, Study Director — The First Affiliated Hospital of Zhengzhou University; Weijun Qin, Study Director — Air Force Medical University of PLA (the Fourth Military Medical University); Lei Li, Study Director — First Affiliated Hospital Xi'an Jiaotong University; Deyi Luo, Study Director — West China School of Medicine of Sichuan University; Zhansong Zhou, Study Director — Southwest Hospital, China; Wei Yu, Study Director — Peking University First Hospital; Jianwei Wang, Study Director — Beijing Jishuitan Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China